CLINICAL TRIAL: NCT05575375
Title: Pilot Randomized Controlled Trial of a Values-Affirmation Intervention Targeting Medication Adherence in Older Adults With Heart Failure
Brief Title: Values-Affirmation + Education Intervention Targeting Medication Adherence in Older Adults With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K23AG061214 (NIH); K23AG061214 (NIH)
Record Dates: First submitted 2022-10-03; First posted 2022-10-12 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Values Affirmation + Usual Care (Experimental)
  Interventions: Behavioral: Values Affirmation + Usual Care
- Usual Care (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Values Affirmation + Usual Care — Participants will engage in a brief values-affirmation exercise to target personal motivation and openness to medication adherence. The interventionist will then review tailored medication education and individual skills training recommendations. The participant's study medication monitoring devices will be labeled with the participants' most important core value(s). Participants will also continue with their usual care.
  Arms: Values Affirmation + Usual Care
Other: Usual Care — Participants will be asked to continue with their usual care (e.g., cardiac rehabilitation, ongoing medical management)
  Arms: Usual Care

SUMMARY:
The goals of this study are to determine the (1) feasibility and (2) acceptability of the study procedures through a pilot randomized controlled trial of a values affirmation intervention targeting medication adherence in adults with heart failure enrolled in cardiac rehabilitation relative to usual care.

DETAILED DESCRIPTION:
Heart failure (HF) represents a significant public health concern. Medication non-adherence is a modifiable contributor to costly hospital readmissions in older adults with HF. Educational interventions improve, but do not eliminate, non-adherence. Values affirmation interventions which invite individuals to reflect on core values may encourage better engagement in health behaviors by increasing the personal relevance of targeted behaviors. This study tests a values-affirmation intervention targeting medication adherence in older adults with HF enrolled in cardiac rehabilitation.

The objective of this study is to examine the feasibility and acceptability of study procedures and the values-affirmation intervention in a pilot randomized controlled trial. Participants will complete a baseline assessment including 30 days of medication monitoring using electronic medication monitoring devices. After the baseline medication monitoring period, participants will be randomly assigned to either the intervention or control condition. Intervention participants will be asked to complete a brief intervention with tailored education relevant to medication information, motivation, and behavioral skills in additional to their usual cardiac rehabilitation care. Control participants will continue with their usual care. Participants will be asked to continue using the medication monitoring devices and to complete a final assessment 30 days later.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure
* Enrolled in cardiac rehabilitation
* Read and understand English

Exclusion Criteria:

* Current participation in another medication-monitoring clinical or research protocol
* New York Heart Association class IV heart failure
* Diagnosis of Alzheimer's, dementia, or severe cognitive impairment indicated on screening
* Current suicidality or psychosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Values Affirmation + Usual Care | Usual Care
Started | 21 | 21
Completed | 21 | 19
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Values Affirmation + Usual Care | Usual Care | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.67 (7.73) | 68.19 (10.54) | 68.43 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 17 | 34
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention and Study Procedures
Description: Participant self-reported satisfaction with intervention content and delivery [intervention group only] and study procedures
Time Frame: Post-test (2-months)
Population: 2 losses to follow-up in intervention group; 1 person did not provide a response to overall acceptability of study procedures in the control group
Measure: Count of Participants; unit: Participants
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 17 | 20
Participants
  Overall Satisfaction with Intervention Content: number analyzed (Participants) | 17 | 0
  Overall Satisfaction with Intervention Content | 17 |
  Overall Satisfaction with Study Procedures | 14 | 17

2. Primary Outcome: Retention
Description: Proportion of enrolled participants who completed the final assessment
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 21 | 21
Participants | 19 | 21

3. Secondary Outcome: Medication Adherence (Electronically Monitored)
Description: Medication adherence will be electronically monitored. Adherence will be calculated as the overall percentage of days in which participants took their medications as prescribed during the monitoring period (30 days for baseline, 30 days post-intervention initiation)
Time Frame: 1 month; calculated as the difference between Baseline and post-test
Population: participants with missing data or data suggestive of non-use (e.g., 3 SDs below mean) excluded
Measure: Mean (Standard Deviation); unit: percentage of days adherent to regimen
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 15 | 14
percentage of days adherent to regimen
  Baseline | 90.27 (14.51) | 88.64 (17.53)
  Posttest: number analyzed (Participants) | 13 | 14
  Posttest | 89.15 (19.45) | 83.14 (19.51)

4. Secondary Outcome: Change in Medication Adherence (Self-report)
Description: Self-reported medication adherence assessed with the Medication Adherence Scale (MAS; Wu et al., 2008). The MAS is a 32-item scale with three subscales - knowledge, attitudes, and barriers-- in addition to items assessing medication-taking behaviors. The 3 subscales are scored by summing items relevant to each subscale. Knowledge subscale scores range from 0 to 30; higher scores indicate greater medication knowledge. Attitudes subscale scores range from 0 to 40, with higher scores indicated report of a more positive attitude towards medication taking. The Barriers subscale scores range from 0 to 110, with higher scores indicated report of more barriers to taking medications as prescribed.
Time Frame: Baseline, post-test (2-months)
Population: 2 participants lost to follow-up at posttest; 2 additional participants missing data at post test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline Attitude subscale | 36.67 (4.55) | 38.05 (2.62)
  Baseline knowledge subscale: number analyzed (Participants) | 20 | 21
  Baseline knowledge subscale | 22.15 (7.14) | 20.76 (8.98)
  baseline barriers subscale | 21.90 (30.05) | 22.00 (32.21)
  posttest Attitude subscale: number analyzed (Participants) | 19 | 21
  posttest Attitude subscale | 38.21 (2.49) | 38.90 (1.26)
  posttest knowledge subscale: number analyzed (Participants) | 19 | 21
  posttest knowledge subscale | 25.16 (4.97) | 22.19 (7.28)
  posttest barriers subscale: number analyzed (Participants) | 17 | 21
  posttest barriers subscale | 16.76 (30.03) | 28.00 (37.92)

5. Secondary Outcome: Medication Adherence (Pill Count)
Description: Pill counts will be conducted on one medication
Time Frame: Baseline, post-test (2-months)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Positive and Negative Affect
Description: Positive and Negative Affect Scale-Short Form (I-PANAS-SF). Two subscales are computed-- the positive affect score and the negative affect score. On both subscales, scores can range from 5 - 25 with higher scores indicating higher positive or negative affect, respectively.
Time Frame: Baseline, post-test (2-months)
Population: 2 participants lost to follow-up and missing posttest data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale
  Positive affect, Baseline | 19.29 (3.88) | 18.57 (5.66)
  Positive Affect, Posttest | 18.74 (4.51) | 19.81 (4.52)
  Negative Affect, Baseline | 7.76 (2.74) | 8.33 (3.26)
  Negative Affect, Posttest: number analyzed (Participants) | 19 | 21
  Negative Affect, Posttest | 7.63 (2.01) | 7.33 (2.46)

7. Other Pre Specified Outcome: Perceived Stress-4
Description: Perceived Stress Scale- 4; total scores range from 0 to 16 with higher scores indicating greater perceived stress over the past month.
Time Frame: Baseline, post-test (2-months)
Population: 2 participants lost to follow-up and missing posttest data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 3.76 (3.42) | 3.86 (3.25)
  Post-Test: number analyzed (Participants) | 21 | 19
  Post-Test | 3.47 (2.74) | 3.00 (3.24)

8. Other Pre Specified Outcome: Medication Self-Efficacy
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions- Managing Medications and Treatment-Short Form 4a Raw scores range from 4 to 20; raw scores were transformed to T-scores with a mean of 50 and a standard deviation of 10. Higher scores reflect higher self-efficacy.
Time Frame: Baseline, post-test (2-months)
Population: missing data for 1 participant at baseline;
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 59.16 (6.16) | 55.97 (6.40)
  posttest: number analyzed (Participants) | 19 | 21
  posttest | 58.45 (5.80) | 58.76 (5.61)

9. Other Pre Specified Outcome: Disease-related Quality of Life
Description: Minnesota Living with Heart Failure Questionnaire; Total scores range from 0 to 105. Higher scores indicate worse health status.
Time Frame: Baseline, post-test (2-months)
Population: 2 participants missing data at post test due to loss to follow-up; 3 additional participants missing data for total score at post test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Values Affirmation + Usual Care | Usual Care
Number analyzed (Participants) | 17 | 21
score on a scale
  Baseline | 26.59 (17.91) | 33.33 (20.41)
  Posttest: number analyzed (Participants) | 16 | 17
  Posttest | 21.50 (26.02) | 27.71 (20.27)

10. Other Pre Specified Outcome: Change in General Quality of Life
Description: EuroQual-5 Dimension (EQ-5D)
Time Frame: Baseline, post-test (2-months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Values Affirmation + Usual Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/21
Other Adverse Events (participants affected / at risk) | 1/21 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Values Affirmation + Usual Care (N=21) | Usual Care (N=21)
myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Values Affirmation + Usual Care (N=21) | Usual Care (N=21)
fall (Musculoskeletal and connective tissue disorders) | 0 | 1
baker's cyst (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05575375/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT05575375/SAP_001.pdf